CLINICAL TRIAL: NCT03317821
Title: PHIL Evaluation in the Endovascular Treatment of Intracranial Dural AVF, a European Multi-center, Observational, Prospective, Single Arm and Open Label Study.
Brief Title: PHIL Evaluation in the Endovascular Treatment of Intracranial Dural AVF
Status: Completed | Type: Observational
Sponsor: Microvention-Terumo, Inc. (Industry)
Collaborators: ClinSearch (Other)
Responsible Party: Sponsor
Other Study IDs: dAVF-Phil Registry
Record Dates: First submitted 2017-10-18; First posted 2017-10-23 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Dural Arteriovenous Fistula
MeSH Terms: conditions — Central Nervous System Vascular Malformations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this study is to demonstrate the safety and efficacy of the PHIL® liquid in endovascular treatment of dural arteriovenous fistula.

DETAILED DESCRIPTION:
This is an European multi-center observational study. Treatments and follow-up visits will be done as per standard of care.

The objective of this study is to evaluate the efficacy and safety of the PHIL® device in the treatment of intracranial dural ArterioVenous Fistula (dAVF). The PHIL® device, a non-adhesive liquid embolic agent, has been CE marked since July 2014. It is intended for use in the embolization of lesions in the peripheral and neurovasculature, including arteriovenous malformations and hypervascular tumors.

All patients with an intracranial dAVF that has not been previously treated and will be treated by embolization with PHIL® are eligible for this study. A maximum of 70 patients will be enrolled in this study in 16 European Institutions.

The expected approximate study duration is 38 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patient or patient's legally authorized representative has received information about data collection and has signed and dated an Informed Consent Form
2. Patient has an intracranial dAVF that can be treated by embolization with PHIL® used with or without other embolization products except other non-adhesive liquid embolic agents (i.e. Squid, Onyx).
3. Patient is at least 18 years of age.

Exclusion Criteria:

1. Patient has multiple dAVFs to be treated.
2. Patient participates in a study evaluating another medical device, procedure, or medication during the course of dAVF treatment and follow-up per the study protocol.
3. Patient does not give consent to the collection and processing of data required for centralized monitoring

3. Any condition that could prevent patient follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patients having an untreated dural arteriovenous fistula requiring treatment will be screened by the investigational sites. Those eligible to be treated with PHIL® will be enrolled after having dated and signed an informed consent form as per appropriate regulation in the participating country.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
Number of adverse events and assessment of neurological status at 1 month after each embolization | 1 month
  Neurological assessment by mRS
Assessment of cure rate and of clinical course of the patient (stable /improvement /deteriorated) | 3-6 months after last embolization
  Cure rate assessment by Angiography

SECONDARY OUTCOMES:
Number of adverse events and assessment of neurological status | 3-6 months after last embolization
  Neurological assessment by mRS
Improvement in the quality of life of the patient and changes in patients symptoms | 3-6 months after last embolization
  Assessed by Quality of Life Questionnaire EQ 5D

CONTACTS AND LOCATIONS:
Locations (16):
- Rigshospitalet University, Copenhagen, Denmark
- France (5):
  - CHU Pellgrin, Bordeaux
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CHU Limoges, Limoges
  - La Fondation Rothschild, Paris
  - Hôpital Pierre Paul Riquet, Toulouse
- Spain (5):
  - Hospital Universitario General de Catalunya, Barcelona
  - Hospital Nuestra Senora del Rosario, Madrid
  - Hospital Regional Universitario Carlos Haya, Málaga
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario Virgen del Rocio, Seville
- Sweden (2):
  - Universitetssjukhus Umea, Umeå
  - Uppsala University, Uppsala
- United Kingdom (3):
  - University Hospital Birmingham, Birmingham
  - Western General Hospital, Edinburgh
  - Charing Cross Hospital, London

IPD SHARING:
Plan to Share IPD: No